CLINICAL TRIAL: NCT02130934
Title: Left Ventricular Strain Assessment Using 3d Cardiac Magnetic Resonance Technique In Asymptomatic Pediatric Patients Who Received Cardiotoxic Chemotherapy
Brief Title: Cardiac 3D MRI in Pediatric Cancer Patients
Status: Withdrawn | Type: Observational
Why Stopped: Slow accrual
Sponsor: Majd Makhoul (Other)
Responsible Party: Sponsor-Investigator, Majd Makhoul, Sponsor/Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 14-0315
Record Dates: First submitted 2014-05-01; First posted 2014-05-06 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Childhood Cancer
Keywords: Childhood cancer; anthracyclines; cardiotoxicity; cardiac MRI; cumulative does of at least 150 mg/m2 of anthracyclines; Ventricular function
MeSH Terms: conditions — Neoplasms; Cardiotoxicity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- childhood cancer survivors: Cardiac 3D MRI
  Interventions: Procedure: Cardiac 3D MRI

INTERVENTIONS:
Procedure: Cardiac 3D MRI

SUMMARY:
This is a non-randomized prospective pilot study in a single academic center with historic controls. This study will compare Cardiac Magnetic Resonance Images (MRI) of patients who have undergone childhood cancer treatment that has cardio-toxic effects to historic controls. The ultimate goal of this study is to develop a safe and effective method for early diagnosis of heart problems in children who are receiving chemotherapy treatments that may be toxic to the heart.

DETAILED DESCRIPTION:
The following tests and procedures will be performed after consent has been obtained. All tests and procedures noted below are being done for the sole purpose of the study:

Visit 1. Subjects will be asked to complete some questionnaires and answer questions regarding smoking status and use of alcohol or smokeless tobacco. We will also gather basic information such as age, height, weight, gender, ethnicity, race, pertinent medical history as well as collect vital sign information (height, weight, blood pressure, heart and respiratory rate.) Next, subjects will undergo a routine transthoracic echocardiogram.

Visit 2. Following the completion of the echocardiogram, and if selected to take part in the study, subjects will be schedule for a cardiac MRI test within a 3 months period.

When subjects come in for Visit 2, they will receive a 12 lead electrocardiograph (ECG) before the cardiac 3D MRI.

All females who are capable of becoming pregnant, except those who are age 11 and under, will then undergo urine pregnancy testing. If it is found that you are pregnant you will not be allowed to be in the study. If the female is under 18 and a positive pregnancy test result is obtained, we will inform both the participant and her parent/guardian.

Subjects may then be placed in a "simulated" MRI to teach them what it will be like to enter the scanner and also train them on how to breathe calmly and regularly during the scan.

Training will involve the use of a PrimeSense 3D sensor, similar to the cameras used in active videogame systems such as the Xbox Kinect, which will generate a 3D picture of their chest as they breathe. Following this training session, subjects will then undergo cardiac 3D MRI. Study participations will end after this visit.

ELIGIBILITY:
Inclusion Criteria:

* Childhood cancer treatment which has been completed
* Received anthracyclines as part of childhood cancer treatment, at least 150 mg/m2 as cumulative dose
* normal left ventricular systolic and diastolic functions on echocardiogram

Exclusion Criteria:

* Ongoing cancer treatment
* Pregnancy
* Inability to undergo a cardiac MRI
* Abnormal ventricular systolic or diastolic function on echocardiogram

Ages: 8 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects will come from the Kentucky Children's Hospital Hematology/Oncology clinic. The study team will ask the subject's primary physician to introduce the study in clinic to any patient who is identified by the study team as meeting the enrollment criteria. If the patient and his/her family are interested in participating, a member of the study team will be notified, and will then consent / assent the patient and family for the study. Patients who wish to consider the study and potentially enroll later will be given contact information to call the study personnel if they wish to enroll later.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Ventricular Function Measurement | Up to 2 years
  Quantify ventricular functional measurements including strain patterns and measurements using offline processing software that Dr. Fornwalt lab has.

CONTACTS AND LOCATIONS:
Overall Officials: Majd Makhoul, MD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - UK Medical Center, Lexington, Kentucky
  - University of Kentucky Medical Center, Lexington, Kentucky